CLINICAL TRIAL: NCT04390074
Title: COVID-19 in the Swedish ICU-cohort: Risk Factors of Critical Care Admission and Intensive Care Mortality
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Center for Clinical Research Dalarna, Sweden (Other)
Responsible Party: Sponsor
Other Study IDs: UTN: U1111-1251-8195
Record Dates: First submitted 2020-05-14; First posted 2020-05-15 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: COVID-19; Critical Illness
MeSH Terms: conditions — COVID-19; Critical Illness | interventions — Critical Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19: Patients with COVID-19 who have received or are receiving Intensive Care in Sweden. Patients are identified in the Swedish Intensive care registry, to which all Swedish intensive care units (ICU) are reporting all intensive care patients.
  Interventions: Other: COVID-19 and Intensive Care
- Control: Age- and sex-matched controls are drawn from all residents of Sweden by Statistics Sweden.

INTERVENTIONS:
Other: COVID-19 and Intensive Care — No intervention, observational.
  Groups: COVID-19

SUMMARY:
The Corona virus disease 2019 (COVID-19) pandemic is currently involving all parts of the world. Several risk factors for critical illness and death from the disease have been proposed. However, the observed associations between different comorbidities and chronic medications have not fully been related to the frequencies of the same comorbidities and chronic medications in age- and sex-matched controls from the general population. This is important since some of the proposed risk factors are very common in the aged who, by age alone, are more prone to a more severe course of the disease.

By combining several registries, we will compare, on several comorbidities such as hypertension and diabetes and several medications such as immunosuppressant drugs and Angiotensin Converting Enzyme (ACE)-inhibitors, the first 2000 cases of COVID-19 patients receiving critical care in Sweden to a set 8000 age- and sex-matched controls.

DETAILED DESCRIPTION:
The COVID-19 pandemic is currently involving all parts of the world. Several risk factors for critical illness and death from the disease have been proposed. However, the observed associations between different comorbidities and chronic medications have not fully been related to the frequencies of the same comorbidities and chronic medications in age- and sex-matched controls from the general population. This is important since some of the proposed risk factors are very common in the aged who, by age alone, are more prone to a more severe course of the disease.

By combining several registries, we will compare, on several comorbidities such as hypertension and diabetes and several medications such as immunosuppressant drugs and ACE-inhibitors, the first 2000 cases of COVID-19 patients receiving critical care in Sweden to a set 8000 age- and sex-matched controls.

Data sources:

Registries of the Swedish board of Health and wellfare:

1. The patient registry containing information including diagnostic codes from all specialized Healthcare contacts in Sweden. Reporting i governed by law.
2. The Swedish Prescribed Drug Register to which all dispensations from pharmacies of prescribed drugs are reported.

Statistics Sweden is the agency responsible for the official population statistics of Sweden. They will draw our controls from the Registry of the total population.

The Swedish Intensive Care Registry (SIR) contains all intensive care episodes in Sweden. They have information on Intensive Care (ICU) admission, diagnoses, interventions and outcomes.

The study design is combined prospective ond retrospective. The data is prospectively collected to the registries but the study protocol is retrospectively designed.

ELIGIBILITY:
Inclusion Criteria:

-Included in the SIR with COVID-19 any time until data acquisition

Exclusion Criteria:

-Age below 18 years.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The SIR is a registry to which all Swedish intensive care units are reporting all intensive care patients. The SIR has a specific part to wich all CIVID-19 related intensive care eposodes are reported. We will include, as cases, all patients, approximally 2000, who have at least one COVID-19 listing in the registry. Statistics Sweden will draw a random sample of age and sex matched controls, 4 per case, from all residents of Sweden, approximately 10 million.
Sampling Method: Probability Sample
Enrollment: 9905 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Chronic medications as risk factor of intensive care for COVID-19 | Drug dispensation within 6 months prior inclusion
  Odds ratio of intensive care treated patients with COVID-19 having ongoing treatment with drugs blocking the Renin-Angiotensin-Aldosterone-System (RAAS), statins, immunosuppressant drugs, oral anticoagulant drugs, oral thrombocyte aggregation inhibitors or antiviral drugs.
Comorbidities as risk factor of intensive care for COVID-19 | 5 years prior to inclusion
  Odds ratio of intensive care treated patients with COVID-19 having been diagnosed with diabetes typ I, diabetes type II, ischemic heart disease, other heart disease, cerebrovascular disease, cancer, chronic renal failure, chronic obstructive pulmonary disease (COPD) asthma, obesity, immunosuppressed disease or systemic inflammatory disease.

SECONDARY OUTCOMES:
Chronic medications as risk factor of death during intensive care for COVID-19 | Drug dispensation within 6 months prior inclusion
  Odds ratio of patients who have died during intensive care with COVID-19 having ongoing treatment with drugs blocking the Renin-Angiotensin-Aldosterone-System (RAAS), statins, immunosuppressant drugs, oral anticoagulant drugs, oral thrombocyte aggregation inhibitors or antiviral drugs.
Comorbidities as risk factor of death during intensive care for COVID-19 | 5 years prior to inclusion
  Odds ratio of patients who have died during intensive care with COVID-19 having been diagnosed with diabetes typ I, diabetes type II, ischemic heart disease, other heart disease, cerebrovascular disease, cancer, chronic renal failure, chronic obstructive pulmonary disease (COPD) asthma, obesity, immunosuppressed disease or systemic inflammatory disease.

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Lipcsey, PhD, Principal Investigator — Uppsala University
Locations (1):
- Björn Ahlström, Falun, Sweden

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD is not allowed under the permission of the ethical review board.